CLINICAL TRIAL: NCT04500587
Title: Phase 1 First in Human Dose-Escalation Study of ZN-d5 as a Single Agent in Subjects With Non-Hodgkin Lymphoma or Acute Myeloid Leukemia
Brief Title: Phase 1 First in Human Study of ZN-d5 as a Single Agent
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: K-Group Alpha, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: ZN-d5-001
Record Dates: First submitted 2020-07-30; First posted 2020-08-05 (Actual); Last update posted 2024-09-19 (Actual); Status verified 2024-09

CONDITIONS: Acute Myeloid Leukemia; Non Hodgkin Lymphoma
Keywords: BCL-2 Inhibitors; BH3 mimetics
MeSH Terms: conditions — Leukemia, Myeloid, Acute; Lymphoma, Non-Hodgkin | interventions — Drug Evaluation

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (2):
- ZN-d5 Single Agent Dose Escalation - NHL (Experimental): Non-Hodgkin Lymphoma
  Interventions: Drug: ZN-d5
- ZN-d5 Single Agent Dose Escalation - AML (Experimental): Acute Myeloid Leukemia
  Interventions: Drug: ZN-d5

INTERVENTIONS:
Drug: ZN-d5 — Oral agent; 25 mg or 100 mg formulation
  Other Names: Study Drug

SUMMARY:
Phase 1 dose escalation study of ZN-d5 in subjects with relapsed or refractory non-Hodgkin lymphoma (NHL) or acute myeloid leukemia (AML).

DETAILED DESCRIPTION:
This is an open-label multicenter Phase 1 dose escalation study evaluating the safety, tolerability, clinical activity, pharmacokinetics and pharmacodynamics of the novel BCL-2 inhibitor ZN-d5 in subjects with (NHL) or (AML) in order to determine the recommended phase 2 dose of ZN-d5.

ELIGIBILITY:
Key Inclusion Criteria:

NHL: relapsed or refractory NHL including DLBCL, FL, MZL, MCL, LCL, LPL and PTC

* Subjects must have received at least 2 prior lines of therapy and have either failed or not be eligible for any available therapies expected to provide clinical benefit and have measurable disease.

AML: Primary, secondary, or treatment-related AML, relapsed or refractory to prior therapy, which may include failure of one cycle of induction therapy.

* White blood cell count < 25 × 109/L. Cytoreduction prior to treatment is acceptable.
* Subjects may not be pregnant and must agree to use an effective method of contraception.
* Eastern Cooperative Oncology Group performance status ≤ 2.
* Estimated life expectancy of at least 12 weeks.
* Adequate hematologic and organ function, including creatinine clearance ≥ 60 mL/min.

Key Exclusion Criteria:

* Recent interventions including major surgery, radiation therapy, stem cell transplant.
* Treatment with anti-neoplastic agents with 5 half-lives.
* Significant unresolved toxicity from prior treatments including active GVHD.
* Active central nervous system disease.
* Clinically substantial myocardial impairment.
* Prior therapy with venetoclax.

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 39 (Actual)
Dates: Start 2020-10-13 (Actual); Primary Completion 2023-12-12 (Actual); Study Completion 2023-12-12 (Actual)

PRIMARY OUTCOMES:
Observed Dose Limiting Toxicities | Through completion of Cycle 1; 1 to 2 months.
  Observed Dose Limiting Toxicities (DLTs) in DLT-evaluable subjects.
Incidence and severity of AEs, graded according to the National Cancer Institute Common Terminology Criteria for Adverse Events, v 5.0 | Through study completion, typically < 12 months
  Safety profile of ZN-d5.

SECONDARY OUTCOMES:
Pharmacokinetic parameters for ZN-d5 - Cmax | approximately 6 months
  Characterize the Pharmacokinetics of ZN-d5 in subjects with NHL and AML using peak plasma concentration (Cmax).
Pharmacokinetic parameters for ZN-d5 - Tmax | approximately 6 months
  Characterize the Pharmacokinetics of ZN-d5 in subjects with NHL and AML using the time to maximum plasma concentration (Tmax).
Pharmacokinetic parameters for ZN-d5 - AUC | approximately 6 months
  Characterize the Pharmacokinetics of ZN-d5 in subjects with NHL and AML using area under the plasma concentration versus time curve (AUC).
For NHL, evaluate response according to the Lugano 2014 classification | Through study completion, typically < 12 months
  Evaluate response according to the Lugano 2014 classification for NHL subjects. The Lugano Classification is based on a 5-point scale for scoring of metabolically active lesions detected by PET-CT in FDG-avid lymphomas, and lesion size for non-FDG-avid tumors. A complete metabolic response would require a score of 1 or 2 on target and non-target lesions and the spleen for high-risk disease, and a score of 1,2, or 3 for low-risk disease. A partial response, no response, or progression would require a score of 4 or 5 for low-risk disease, and a score of 3, 4, or 5 for high-risk disease.
For AML, remission rate based on European LeukemiaNet 2017 criteria | Through study completion, typically < 12 months
  Evaluate remission rate according to the European LeukemiaNet 2017 criteria (Overall Response Rate (ORR) defined as Complete Remission (CR) + CR with incomplete hematologic recovery (CRi) + Morphologic Leukemia-Free State (MLFS) + Partial Remission (PR)) for AML subjects.
For AML, duration of remission based on European LeukemiaNet 2017 criteria | Through study completion, typically < 12 months
  Evaluate duration of remission according to the European LeukemiaNet 2017 criteria.

CONTACTS AND LOCATIONS:
Overall Officials: K-Group Alpha Inc. /a subsidiary of Zentalis Pharmaceuticals, Study Director — K-Group Alpha, Inc., a wholly owned subsidiary of Zentalis Pharmaceuticals, Inc.
Locations (14):
- Australia (4):
  - Site 2708, Darlinghurst, New South Wales
  - Site 2704, Liverpool, New South Wales
  - Site 2710, Kurralta Park, South Australia
  - Site 2709, Hobart, Tasmania
- Bulgaria (2):
  - Site 1202, Sofia
  - Site 1201, Varna
- Site 3201, Zagreb, Croatia
- Site 2403, Gdansk, Poland
- South Korea (2):
  - Site 2901, Pusan
  - Site 2903, Seoul
- Spain (3):
  - Site 3001, Barcelona
  - Site 3005, Bilbao
  - Site 3003, Valencia
- Site 2001, Kiev, Ukraine

IPD SHARING:
Plan to Share IPD: No